CLINICAL TRIAL: NCT00999947
Title: Genetic Study of Arrhythmogenic Right Ventricular Dysplasia/Cardiomyopathy
Brief Title: Arrhythmogenic Right Ventricular Dysplasia/Cardiomyopathy
Acronym: DVDA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P051067
Record Dates: First submitted 2009-09-29; First posted 2009-10-22 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2012-10

CONDITIONS: Cardiomyopathy; Arrhythmogenic Right Ventricular Dysplasia
Keywords: genetics; mutation screening; phenotype-genotype analysis; desmosomal genes
MeSH Terms: conditions — Cardiomyopathies; Arrhythmogenic Right Ventricular Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this trial is to study the genetic and phenotypic aspects of Arrhythmogenic Right Ventricular Dysplasia/Cardiomyopathy (ARVD/C), and determine the impact of genetic testing in clinical practice.

DETAILED DESCRIPTION:
Arrhythmogenic right ventricular dysplasia/cardiomyopathy (ARVD/ARVC), is an inherited myocardial disease that predominantly affects the right ventricle (RV) and the estimated prevalence in the general population ranges from 1 to 5 in 1000. It is characterized histopathologically by fibro-fatty myocardial replacement and clinically by ventricular arrhythmia that may lead to sudden death, especially in young people and athletes. Clinical diagnosis is based on diagnostic criteria proposed by the International Task Force of the European Society of Cardiology and International Society and Federation of Cardiology (Task Force 1994), but is often difficult due to a broad spectrum of clinical features and a lond period of concealed cardiac expression, with delayed diagnosis.

ARVC/D is familial in 30 to 50% and is typically transmitted as an autosomal dominant trait with variable penetrance. In the past years, the identification of causative mutations in plakoglobin (JUP), desmoplakin (DSP), plakophilin-2 (PKP2), desmoglein-2 (DSG2), desmocollin-2 (DSC2) has fostered the view that ARVC/D is a disorder of the desmosome and provided new insight into its pathogenesis.

The major recent advance in the molecular genetics of ARVD/C might lead to important clinical impact through early and correct diagnosis in patients and relatives, and through potential genotype-phenotype correlations. This key-issue requires first to clarify the optimal molecular strategy, and its efficiency. Such a systematic, detailed and comprehensive mutation screening study is not available until now.

Aim:

Study the genetic and phenotypic aspects of Arrhythmogenic Right Ventricular Dysplasia/Cardiomyopathy (ARVD/C), and determine the impact of genetic testing in clinical practice.

Methods:

The study was approved by the Pitié-Salpétriêre Hospital ethical committee (CPPRB) and written informed consent was obtained from all participating individuals, recruited in France.

A cohort of 100 unrelated patients with ARVD/C will be recruited. Clinical evaluation will include clinical history, family history, blood sample for DNA analysis 12-lead ECG, signal-average ECG, 24-hour ambulatory ECG, transthoracic echocardiography, MRI and/or radionuclide scintigraphy, and contrast angiography when possible. A clinical diagnosis of ARVD/C is made according to the established European Society of Cardiology / International Society and Federation of Cardiology Task Force major and minor criteria (Task Force 1994).

All available relatives will be proposed for enrollment in the study with blood sample for DNA analysis and non invasive cardiac examination, including 12-lead ECG, signal-average ECG, and transthoracic echocardiography.

Mutational analysis of the five genes encoding desmosomal genes will be performed in all index cases (in plakoglobin, desmoplakin, plakophilin-2, desmoglein-2, desmocollin-2). When mutations will be identified, available relatives will be analysed. In index cases without desmosomal mutation, additional analyses will be performed according to a candidate gene strategy and, when possible, through a genome wide approach and linkage analyses.

Expected results:

Determine the genetic origin in patients with ARVD/C whatever the familial context.

Determine a molecular strategy for routine genetic testing. Determine the impact of genetic testing as a diagnostic test in patients and relatives.

Determine the impact of genetics as a prognostic tool, through phenotype-genotype analyses.

Determine the natural evolution of the disease in relatives, and the penetrance.

ELIGIBILITY:
Inclusion Criteria:

* Patient with DVDA diagnostic confirmed
* Acceptance even follow-up
* Informed consent

Exclusion Criteria:

* Impossible to understand the notice information about study
* Not affiliated with social protection

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Unrelated patients with ARVD/C. A clinical diagnosis of ARVD/C is made according to the established European Society of Cardiology / International Society and Federation of Cardiology Task Force major and minor criteria (Task Force 1994)
  + All available relatives will be proposed for enrollement in the study
Sampling Method: Non-Probability Sample
Enrollment: 351 (Actual)
Dates: Start 2006-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Determine the genetic origin in patients with ARVD/C whatever the familial context | at inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Charron, MD, PhD, Principal Investigator — Pitié-Salpêtrière Hospital
Locations (1):
- Pitié-Salpêtrière Hospital, Paris, France